CLINICAL TRIAL: NCT05148039
Title: Comprehensive Assessment of Nutrition & Dietary Intervention in Hypermobile Ehlers Danlos Syndrome (hEDS/HSD): a Personalised Approach: Phase 2 & 3
Brief Title: Comprehensive Assessment of Nutrition and Dietary Intervention in Hypermobile Ehlers Danlos Syndrome
Acronym: CANDI-hEDS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 306930
Record Dates: First submitted 2021-11-16; First posted 2021-12-08 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Hypermobile Ehlers-Danlos Syndrome; Irritable Bowel Syndrome; Functional Gastrointestinal Disorders
Keywords: Nutrition; Diet
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Tertiary clinic versus a selective community cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community cohort (Active Comparator): Participants from the Ehlers Danlos UK society community who low diet quality
  Interventions: Behavioral: Dietician advice
- Clinic cohort (Active Comparator): Participants from a Tertiary Neurogastroenterology clinic who have low die quality
  Interventions: Behavioral: Dietician advice

INTERVENTIONS:
Behavioral: Dietician advice — Personalised dietetic advice

SUMMARY:
This study involves a comprehensive nutritional assessment of hEDS participants who have functional gastrointestinal disorders and dietary intervention to broaden their food choices and nutritional intake.

DETAILED DESCRIPTION:
The impact of diet on symptoms in patients with Hypermobile Ehlers Danlos Syndrome (hEDS/HSD) is widely recognised yet poorly understood. The investigators aim is to assess existing dietary patterns and nutritional status in hEDS/HSD as well as pilot a personalised dietary strategy to optimise nutrition. Participants recruited from EDS UK and a tertiary Neurogastroenterology clinic at the Royal London Hospital will undergo comprehensive nutritional assessment and blood tests. The investigators will then undertake a feasibility study of personalised dietary intervention in select cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Have completed Phase I of the CANDI-hEDS study
* Diagnosis of hEDS / HSD according to physical examination and history taking
* Diagnosis of Functional Dyspepsia and / or Irritable Bowel Syndrome according to Rome IV criteria
* Able and willing to give informed consent
* Access to video conferencing and a smart phone device
* Able to travel to the Wingate Institute

Exclusion Criteria:

* Dependent upon artificial feeding (parenteral and enteral)
* Structural gastrointestinal disease
* Any chronic health condition which already requires a restricted diet e.g. diabetes mellitus
* Functional vomiting disorder with associated weight loss
* Multiple Type I hypersensitivity reactions to food groups (i.e. anaphylaxis, urticaria, respiratory symptoms or positive RAST tests).
* Previous or current severe mental health disorder (e.g. severe depression with suicidal ideation)
* Previous or current eating disorder
* Positive screen for avoidant restrictive food intake disorder (ARFID)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Number of patients | 3 months
  Number of patients who adhere to dietary recommendations based on acceptability of intervention and ease of delivery.

SECONDARY OUTCOMES:
United Kingdom Diet Quality Index as calculated by the Scottish Collaborative Group Food Frequency Questionnaire (SCG FFQ) | 3 months
  170- item semi-quantitative questionnaire, designed to assess the habitual diet of medium to large sized populations during the previous 3 months (higher score means better diet quality)
Gastrointestinal Symptom Rating Scale (GSRS) | 3 months
  13-item questionnaire assessing gastrointestinal symptoms across five domains (pain, bloating, constipation, diarrhoea and satiety) over a period of one week. (min:0 max: 7, higher score means worse symptoms)
Hospital Anxiety and Depression Scale (HADS) | 3 months
  14-item scale assessing symptoms of either anxiety or depression (min: 0 max: 21, higher score means worse anxiety or depression)
Visceral Sensitivity Index (VSI) | 3 months
  15-item measurement of gastrointestinal-specific anxiety (min: 0 max: 75, higher score means worse gastrointestinal specific anxiety)
Patient Health Questionnaire-15 (PHQ-15) | 3 months
  15-item questionnaire to assess the domain of somatic symptoms (min: 0 max: 30, higher score means worse somatic symptoms)
Composite Autonomic Symptom Score (COMPASS-31) | 3 months
  31-item score to assess for symptoms of autonomic nervous system disturbance (min: 0 max 100, higher score means worse autonomic symptoms)
Short Form 6D version 2 (SF-6Dv2) | 3 months
  6-item questionnaire to assess impact of physical symptoms on daily functioning and quality of life (ranges from 1 (full health) to -0.574 (worst health); 0 (death))
Resource Use Questionnaire | 3 months
  16-item questionnaire to assess healthcare and health product utilisation over the preceding 3 months (no minimum / maximum, no score)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Marys University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided